CLINICAL TRIAL: NCT05162209
Title: Effects Of Synbiotic Supplementation On Anthropometric Measurements, Glucose Metabolism, Lipid Parameters And Intestinal Microbiota Composition In Children With Exogenous Obesity: (Probesity-2 Study)
Brief Title: PROBESITY-2: Synbiotics in Pediatric Obesity
Acronym: PROBESITY-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PROB2018
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Obesity, Childhood; Obesity, Adolescent
Keywords: Obesity; Synbiotic; Microbiota; Microbiome
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled clinical study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Experimental): Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium bifidum, Bifidobacterium longum, Enterococcus faecium (total 2.5 x10 9CFU/sachet), fructooligosaccharydes (FOS) 625 mg, oral sachet daily, for 12 weeks
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): Oral sachet daily for 12 weeks
  Interventions: Dietary Supplement: Synbiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic — Oral sachet, for 12 weeks

SUMMARY:
The global obesity epidemic presents an unprecedented challenge to the public health worldwide. The factors associated with obesity are complex, and include health behaviours, such as eating habits and daily physical activity, and broader social, environmental and biological determinants that influence these health behaviours. The intestinal microbiota has several beneficial functions related to host health and accumulating evidence indicates that the gut microbiota plays a significant role in the development of obesity, obesity-associated inflammation and insulin resistance. Differences in community composition, functional genes and metabolic activities of the gut microbiota appear to distinguish lean vs obese individuals, suggesting that gut 'dysbiosis' contributes to the development of obesity and/or its complications. Recent studies have suggested some beneficial effects of probiotics and/or prebiotics on obesity and metabolic syndrome in adults; such experience is limited in children and adolescents. There are limited information about the synbiotics in children and adolescent with obesity.The mechanism of action of probotics on obesity are scarce and microbiota restoration/reshaping might be the one. The objective of this study tested the effects of a multispecies synbiotic on anthropometric measurement, glucose metabolism, lipid parameters and intestinal microbiota in children with exogenous obesity.

DETAILED DESCRIPTION:
The global obesity epidemic presents an unprecedented challenge to the public health worldwide. The factors associated with obesity are complex, and include health behaviours, such as eating habits and daily physical activity, and broader social, environmental and biological determinants that influence these health behaviours. The intestinal microbiota has several beneficial functions related to host health and accumulating evidence indicates that the gut microbiota plays a significant role in the development of obesity, obesity-associated inflammation and insulin resistance. Differences in community composition, functional genes and metabolic activities of the gut microbiota appear to distinguish lean vs obese individuals, suggesting that gut 'dysbiosis' contributes to the development of obesity and/or its complications. Recent studies have suggested some beneficial effects of probiotics and/or prebiotics on obesity and metabolic syndrome in adults; such experience is limited in children and adolescents. There are limited information about the synbiotics in children and adolescent with obesity.The mechanism of action of probotics on obesity are scarce and microbiota restoration/reshaping might be the one. The objective of this study tested the effects of a multispecies synbiotic on anthropometric measurement, glucose metabolism, lipid parameters and intestinal microbiota in children with exogenous obesity.

This is a randomized, double-blind, placebo-controlled clinical study with 61 children, aged between 8 to 17 years-old, with exogenous obesity which received a daily dose of a multispecies symbiotic formulation or a placebo for 12 weeks. At entry, the anthropometric measures included weight, height, waist and hip circumference were recorded. Waist circumference to height ratio, waist circumference to hip circumference ratio and body mass index (BMI) was calculated. Venous blood samples were drawn after a minimum 8 hours fasting for measures including serum glucose, insulin, total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides, C-reactive protein (CRP), erythrocyte sedimentation rate; at admission and 12 weeks later. Both groups were treated with a standard diet and increased physical activity. Patients were randomly allocated into two groups in a ratio of 1:1. Randomization with permutated blocks was done using the online software tool. First group received a daily synbiotic supplementation which consisted of a daily probiotic mixture including Lactobacillus acidophilus), Lactobacillus rhamnosus, Bifidobacterium bifidum, Bifidobacterium longum, Enterococcus faecium (total 2.5 x109CFU/sachet), fructooligosaccharydes (FOS) 625 mg, lactulose 400 mg, vitamin A (6 mg), B1 (1.8 mg), B2 (1.6 mg), B6 (2.4 mg), E (30 mg), C (75 mg) for 12 weeks. Second group received placebo for 12 weeks. Each visit (Day 0 and 12 weeks later), stool samples were also collected. The V3 and V4 regions of the 16S rRNA gene were amplified following the 16S Metagenomic Sequencing Library Preparation. The primary end point of this study was to evaluate the effect of the multispecies synbiotic would on weight loss (reduction as percentage for weight and body mass index). Secondary endpoints were the evolution of the other anthropometeic measurements, glucose and lipid metabolism and intestinal microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents
* Aged between 8 to 17 years old with exogenous obesity

Exclusion Criteria:

* Children and adolescents with endogenous obesity
* Children with adolescents with a history of gastrointestinal surgery
* Children with adolescents with chronic intestinal disorders including inflammatory bowel disease
* Children receiving probiotics and /or antibiotics 8 weeks prior this study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change as percentage for weight and body mass index. | 12 weeks
  % reduction comparing to baseline

SECONDARY OUTCOMES:
Change as percentage of anthropometric measurement | 12 weeks
  Waist circumference, hip circumference, waist/hip ratio, waist/height ratio
Change of glucose metabolism | 12 weeks
  Reduction as percentage of HOMA-IR
Change of lipid metabolism | 12 weeks
  Serum total cholesterol, LDL-C, HDL-C, serum triglyceride
Change of Intestinal microbiota composition | 12 weeks
  Change of predominant bacterial genera

CONTACTS AND LOCATIONS:
Overall Officials: Ener C Dinleyici, MD, Principal Investigator — Eskisehir Osmangazi University Faculty of Medicine
Locations (1):
- Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilic Yildirim G, Dinleyici M, Vandenplas Y, Dinleyici EC. Effects of synbiotic supplementation on intestinal microbiota composition in children and adolescents with exogenous obesity: (Probesity-2 trial). Gut Pathog. 2023 Jul 21;15(1):36. doi: 10.1186/s13099-023-00563-y. PMID 37474971
- [Derived] Kilic Yildirim G, Dinleyici M, Vandenplas Y, Dinleyici EC. Effects of Multispecies Synbiotic Supplementation on Anthropometric Measurements, Glucose and Lipid Parameters in Children With Exogenous Obesity: A Randomized, Double Blind, Placebo-Controlled Clinical Trial (Probesity-2 Trial). Front Nutr. 2022 Jul 1;9:898037. doi: 10.3389/fnut.2022.898037. eCollection 2022. PMID 35845797